CLINICAL TRIAL: NCT03913507
Title: Efficacy of a New Sweat Collection Support: Impact on Neonatal Screening and Early Treatment of Cystic Fibrosis
Acronym: MACRODUCT-3710
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/14JUI/253
Record Dates: First submitted 2019-02-21; First posted 2019-04-12 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis Children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- one group : patients with suspicion of cystic fibrosis (Experimental)
  Interventions: Device: Macroduct® Advanced Model 3710 SYS, Wescor

INTERVENTIONS:
Device: Macroduct® Advanced Model 3710 SYS, Wescor — for each subject, both methods will be tested in order to compare the efficacy of the new sweat collection method (Macroduct® Advanced Model 3710 SYS, Wescor) to the method currently used in clinical routine.

SUMMARY:
In nearly 25% of children under 3 months, the sweat test produces a quantity of sweat that does not meet international recommendations and is insufficient to allow reliable and reproducible biological analyzes in the sweat collected. In children between 3 and 12 months, this rate is about 10% when it should not exceed 5%. Insufficient amount of sweat prevents confirmation or reversal of the early diagnosis of cystic fibrosis and early treatment before irreversible complications of the disease.

In this trial, a new support of sweat collection (Macroduct® Advanced Model 3710 Sweat Collection System, Wescor) will be tested with the goal to increase the amount of sweat collected during the sweat test, in comparison with the clinical routine method.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged of 2 days to 12 months
* Indication of a sweat test prescribed by a clinician in a context of neonatal screening
* Clinically stable
* Well hydrated
* Not under treatment with mineralocorticoids

Exclusion Criteria:

* Subjects weighing less than 2 kg
* Subjects less than 48 hours old
* Presence of an acute infectious condition
* Presence of mineralocorticoid treatment

Ages: 2 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2018-07-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-22 (Actual)

PRIMARY OUTCOMES:
chloride concentration | day 1
  The volume and the chloride concentration will be analyzed for each subject.

SECONDARY OUTCOMES:
sweat | day 1
  sweat collected with sweat collection method (Macroduct® Advanced) Model 3710 SYS, Wescor) compared with that currently used in clinical routine.
  The effectiveness criterion of the new Macroduct Advanced collector will be defined as follows: the new device tested will be considered effective if the insufficient amount of sweat levels obtained are smaller or equal to those recommended, i.e. if it is lower than 10% in children under 3 months and below 5% in children between 3 and 12 months.
  The insufficient amount of sweat rates will be compared between the two methods.

CONTACTS AND LOCATIONS:
Overall Officials: Teresinha Leal, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires St Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided